CLINICAL TRIAL: NCT06191211
Title: Can Routine Consultations be Used to Reduce COVID-19 Misinformation and Increase Vaccine Uptake? An Experimental Study in Ghana
Brief Title: Can Doctors Reduce COVID-19 Misinformation and Increase Vaccine Uptake in Ghana? A Cluster-randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: Innovations for Poverty Action (Other); Ghana Health Services (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 214743
Record Dates: First submitted 2023-12-29; First posted 2024-01-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: Vaccination Hesitancy; Communication
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy; Communication | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Standard of care - no engagement or communication skills training for first-line providers.
- Doctors Light Communication (Active Comparator): In facilities randomised to this group, all front-line health workers receiving patients in outpatient consultations over the trial duration will be asked to encourage eligible patients to get vaccinated or receive a booster of the Covid-19 vaccine.
  At the start of the intervention period, all facilities will receive a visit from the District office of the Ghana Health Service. The visit will (1) remind them of the importance of covid19 vaccination to all consulting staff; (2) ask all consulting staff to have discussions with patients about Covid19 vaccination during routine consultations and (3) provide a simple tracking sheet to be used by consulting staff to record these consultations.
  Interventions: Behavioral: Facility engagement
- Doctors Enhanced Communication (Experimental): In addition to facility engagement described in the "Doctor light communication" group, five front-line health workers from each of the facilities in the treatment group will be invited to take part in a training providing information and developing specific communication skills to encourage patients to get vaccinated. The communication skills are based on principles rooted in Motivational Interviewing (MI) and have been used in Ghana to address vaccine hesitancy.
  Interventions: Behavioral: Motivational Interviewing, AIMS; Behavioral: Facility engagement

INTERVENTIONS:
Behavioral: Motivational Interviewing, AIMS — Motivational interviewing (MI). MI is an approach to patient engagement which promotes a collaborative conversation style for strengthening a person's own motivation and commitment to change. With MI, the doctor facilitates patient exploration of potential reasons for behaviour change in the context of what is important to the patient, rather than the physician directly telling the patient what to do. MI has been found more effective than other approaches to patient engagement and health behaviour change and can be effectively taught to primary care providers.
  Arms: Doctors Enhanced Communication
Behavioral: Facility engagement — A letter to the facility from the local health officials; a meeting with the facility manager and health staff to formally announce that we would like providers to encourage COVID-19 vaccinations; deploying a tracking sheet for vaccinations.
  Arms: Doctors Enhanced Communication; Doctors Light Communication

SUMMARY:
Whilst Ghana was one of the first countries to start vaccinating its population against COVID-19, less than 30% of the population was fully vaccinated at the end of 2022. To improve COVID-19 vaccine uptake, the government has so far relied on two strategies: sensitization in communities and specific national vaccination days. Against the backdrop of strict budget constraints and the return to normalcy in health-seeking behaviours, the investigators aim to test the effectiveness of leveraging interactions of patients with the healthcare system to reduce misinformation and increase vaccination. The investigators collaborate with the Ghana Health Service to offer vaccination as a default option during routine consultations. To dispel information and encourage vaccination uptake effectively, the investigators test two interventions designed to encourage and equip front-line providers with skills to discuss COVID-19 vaccination with patients. The study evaluates the effect of the two interventions in a cluster-randomised trial where the investigators allocate 120 facilities to one of three groups: a control group where providers are not asked to offer COVID-19 vaccines; a light engagement group, where providers receive information about COVID-19 and vaccines and a light-touch vaccine monitoring device is deployed in their facility, and a communication skills building group, where providers receive all the elements of the light intervention, plus training in motivational engagement techniques to encourage vaccination. The primary outcome will be vaccination uptake and intentions. The study will also evaluate the impact of the intervention on patients' knowledge, beliefs and satisfaction. The investigators will track the effectiveness of the training on providers as well as the extent to which they apply their training to actual practice. Results will contribute to a nascent evidence base on potential ways to encourage adult vaccination during routine consultations.

ELIGIBILITY:
Inclusion Criteria:

* Mentally sound adults who are aged 16 years and above
* Presenting at the health centre on the day of surveys

Exclusion Criteria:

* Received a COVID-19 vaccination dose within last 6 months, or received 2 or more doses
* Have fever, chills, or are experiencing severe pain

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
COVID-19 vaccination uptake rates in the health centre | 8 weeks
Proportion of patients who intend to get vaccinated | Immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ghana Health Service, Accra, Greater Accra Region, Ghana

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share a complete dataset at the individual-level containing all primary and secondary study outcomes, any other variables used in the analysis, and treatment assignments. Data will be anonymised to ensure no participants can be personally identified (directly or indirectly)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available permanently. They will become available along with the publication of the study in a journal, as we will provide a replication package as part of the publication.